CLINICAL TRIAL: NCT01122199
Title: Phase I Study of mTOR Inhibitor RAD001 in Combination With IGF-1R Inhibitor AMG479 for Patients With Advanced Solid Tumors
Brief Title: Study of RAD001 + AMG479 for Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shadia Jalal (Other)
Collaborators: Amgen (Industry); Novartis (Industry)
Responsible Party: Sponsor-Investigator, Shadia Jalal, Assistant Professor of Medicine, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1002-16; IUCRO-0287
Record Dates: First submitted 2010-05-07; First posted 2010-05-13 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Neoplasm Metastases
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Everolimus; ganitumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label (Experimental): RAD001+ AMG479
  Interventions: Drug: RAD001 + AMG479

INTERVENTIONS:
Drug: RAD001 + AMG479 — Escalating doses of RAD001 + AMG479. Starting cohort will be 5 mg RAD001 once daily, continuous + AMG479 12 mg/kg on Day 1 and 15 of each 28 day cycle.
  Other Names: everolimus + ganitumab

SUMMARY:
The purpose of this study is to test the safety of the combination of two drugs called RAD001 and AMG479. This study will see what effects (good and bad) RAD001 and AMG479 have on cancer. This study will also find the highest doses of RAD001 and AMG479 that can be given without causing severe side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated (MTD) and recommended Phase II doses for AMG479 (ganitumab) and RAD001 (everolimus) in patients with refractory solid tumors.

II. To determine the safety and toxicity of AMG479 and RAD001.

SECONDARY OBJECTIVES:

I. To determine preliminary antitumor efficacy of AMG479 and RAD001 in solid tumors: response and stable disease rates, duration of response and of stable disease, time to progression (TTP) and overall survival (OS).

II. For all patients, to analyze tumor and blood samples for pharmacodynamic biomarkers related to IGF-1R and mTOR signaling: pAkt, pS6, p-4EBP1, PTEN, IGF-1, IGF-2, pIGF-1R and IGFBP3 and correlate with response and stable disease.

III. For all patients, to analyze the pharmacokinetic profile (PK) for RAD001 and AMG479, and correlate with response/stable disease and pharmacodynamic markers.

IV. To evaluate the effects of RAD001 on AMG 479 pharmacokinetics.

OUTLINE: This is a dose-escalation study.

Patients receive everolimus orally (PO) once daily (QD) on days 1-28 (days 1-7 and 16-28 of course 1 only) and ganitumab intravenously (IV) over 60 minutes on days 1 and 15 (day 15 of course 1 only). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at day 30, every 3 months for 2 years from registration for study treatment, every 6 months for years 3-5, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of metastatic solid tumor refractory to standard therapies, or for which no standard therapies are available.
* Patients in the expansion cohort must have a measurable site of disease according to RECIST (v 1.0)
* Laboratory values must be obtained within protocol limits and obtained within 14 days prior to registration
* Patients must have disease which is not amenable to potentially curative surgical resection of metastatic disease (curative metastasectomy).
* Must be willing to provide metastatic tissue biopsy samples (may be paraffin embedded) at baseline
* Must be willing to undergo a metastatic tissue biopsy after 2 cycles of therapy to perform pharmacodynamic research biomarkers testing.
* Subjects must be willing and able to abstain from using strong or moderate CYP3A4 inhibitors or inducers during the study period.

Exclusion Criteria:

* No symptomatic brain metastasis
* No prior treatment with an mTOR inhibitor or with an IGF-1R inhibitor
* No known history of diabetes mellitus
* No thrombosis or vascular ischemic events within the last twelve months
* No chronic treatment with systemic steroids or another immunosuppressive agent
* No active bleeding or a pathological condition that is associated with a high risk of bleeding
* No known history of HIV seropositivity
* No known history of Hepatitis B or Hepatitis C seropositivity
* No known hypersensitivity to AMG 479, RAD001 (everolimus), other rapamycins (sirolimus, temsirolimus), or to its excipients
* No planned immunization with attenuated live viruses during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-05-14 (Actual); Primary Completion 2015-01-19 (Actual); Study Completion 2015-01-19 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated (MTD) and recommended Phase II doses for AMG479 and RAD001 in patients with refractory solid tumors | 1 year
To evaluate the grade and severity of adverse events as a measure of safety and toxicity | 2 years

SECONDARY OUTCOMES:
To determine preliminary antitumor efficacy of AMG479 and RAD001 in solid tumors | 5-10 years
  response and stable disease rates, duration of response and of stable disease, time to progression (TTP) and overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Shadia I Jalal, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States